CLINICAL TRIAL: NCT04601571
Title: Confirming Feeding Tube Position Using the CORTRAK Enteral Access System
Brief Title: Confirming Feeding Tube Position Using CORTRAK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite the study being in active enrollment since 2020, the research staff has not been available to enroll patients because of lack of trained nursing staff.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20200625H
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: A non-inferior cohort study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Feeding Tube Placement using CORTRAK stylet (Active Comparator): Subjects will already have a feeding tube placed and are undergoing X-rays for placement confirmation.
  Interventions: Device: CORTRAK Stylet
- Feeding Tube Placement using X-Ray (No Intervention): Routine X-ray is used to confirm feeding tube placement

INTERVENTIONS:
Device: CORTRAK Stylet — The stylet is a component of the CORTRAK feeding tube system used to confirm the correct placement of the feeding tube
  Other Names: Feeding tube stylet
  Arms: Feeding Tube Placement using CORTRAK stylet

SUMMARY:
This study will compare the accuracy of the CORTRAK enteral access system (CEAS) to x-ray for the determination of feeding tube position within the abdomen.

DETAILED DESCRIPTION:
In the inpatient pediatric care area (PICU, PCCU, PIMU, ACU), when an x-ray is performed for any reason and a patient has a CORTRAK feeding tube, a provider from the research team will re-insert the small, individualized, flexible stylet back into the patient's feeding tube and document the position of the tube on the CORTRAK display monitor. The x-ray will be obtained by current standard of care and the tube location on x-ray will be compared to the tube location on the CORTRAK monitor. The x-ray will only be obtained as part of the routine care decided by the medical team, the patient will not receive any additional x-rays for this study.

ELIGIBILITY:
Inclusion Criteria:

* CORTRAK feeding tube placed as part of clinical care
* Getting xray for any reason
* CORTRAK Stylet available in the room
* Pediatric patients (Aged 17 or younger)

Exclusion Criteria:

-CORTRAK Stylet has been misplaced

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Confirmation of correct placement of the Feeding tube | Baseline to removal of feeding tube (on average 10-14 days)
  An x-ray will be obtained first as per standard of care and within 4 hours of the x-ray, the research procedure will occur. Following slow and careful removal of the stylet, the research team member will ensure there has been no movement of the feeding tube per the depth indicators on the outside of the tube. The location of the tube as it appears on the CORTRAK monitor will be documented and the location of the tube on x-ray will be documented. This will be reported as number of times that the tube is correctly placed.

SECONDARY OUTCOMES:
Number of Radiographs required for placement | Baseline to removal of feeding tube (on average 10-14 days)
  Count of radiographs used to ensure correct placement of enteral feeding tube

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Meyer, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- University Health Systems Hospital, San Antonio, Texas, United States